CLINICAL TRIAL: NCT04044287
Title: Sublingual Misoprostol and Routine Third Stage Prophylaxis for the Prevention of Postpartum Haemorrhage: A Randomised Controlled Clinical Trial.
Brief Title: Misoprostol in the Prevention of Postpartum Haemorrhage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECP 200 11/12
Record Dates: First submitted 2019-04-04; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2018-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): 200 micrograms of Misoprostol applied sublingually together with standard parenteral oxytocic therapy
  Interventions: Drug: 200 micrograms of misoprostol
- Placebo (Placebo Comparator): 200 micrograms of powdered placebo applied sublingually together with standard parenteral oxytocic therapy micrograms of misoprostol
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: 200 micrograms of misoprostol — 200 micrograms of powdered misoprostol applied sublingually together with standard parenteral oxytocic therapy
  Arms: Intervention
Drug: Placebo Oral Tablet — 200 micrograms of powdered placebo applied sublingually together with standard parenteral oxytocic therapy
  Arms: Placebo

SUMMARY:
Postpartum haemorrhage is a major contributor to maternal mortality in the developing world. The incidence is between 5 and 12% in Jamaica and varies depending on the route of delivery. Misoprostol is a uterotonic agent which has the potential to augment the effects of the standard parenteral oxytocic agents used as best practice in the active management of the third stage of labour, thereby reducing the risk of postpartum haemorrhage and its attendant complications.

The Aim of the study is twofold: to show that this additive effect translates to a reduced postpartum haemorrhage rate and secondly to demonstrate reduced side effects of misoprostol resulting from the lower dose and the powdered sublingual administration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to the labour wards at University Hospital of the West Indies (UHWI) and Victoria Jubilee Hospital (VJH) undergoing a vaginal delivery
* Consent given to participate in the study

Exclusion Criteria:

* Women undergoing caesarean section
* Gestational age less than 28 weeks
* Any severe allergic conditions
* Severe asthmatics
* Age <16 years
* Temperature >38 degrees Celsius
* Women not wishing to consent to join the study

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1496 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume of blood loss at the time of delivery | 24 hours
  Volume (ml) of blood loss at the time of delivery will be measured using an under-buttock collection drape

SECONDARY OUTCOMES:
Comparison of blood loss between intervention and control group | 24 hours
  Volume of blood loss at delivery in the control group.
Measurement of Haematological indices (Haemoglobin level) | 24 hours
  Measurement of haemoglobin level (g/dl) in blood samples obtained on admission in labour compared to 24 hours postpartum
Comparison of Haematological indices (Packed Cell Volume, PCV) | 24 hours
  Measurement of the PCV (%) in blood samples obtained on admission in labour compared to 24 hours postpartum
Measurement of Electrolytes (Sodium) | 24 hours
  Blood concentration of sodium (mmol/L) will be measured on admission in labour compared to 24 hours postpartum
Measurement of Electrolytes (Potassium) | 24 hours
  Blood concentration of potassium (mmol/L) will be measured on admission in labour compared to 24 hours postpartum
Measurement of Electrolytes (Chloride) | 24 hours
  Blood concentration of chloride (mmol/L) will be measured on admission in labour compared to 24 hours postpartum
Measurement of Electrolytes (Bicarbonate) | 24 hours
  Blood concentration of bicarbonate (mmol/L) will be measured on admission in labour compared to 24 hours postpartum
Cardiovascular instability - Frequency of hypotension as a complication of bleeding | 24 hours
  Presence of hypotension will be assessed as cardiovascular instability due to a complication of bleeding in each participant on admission in labour compared to 24 hours postpartum
Cardiovascular instability - Frequency of tachycardia as a complication of bleeding | 24 hours
  Presence of tachycardia will be assessed as cardiovascular instability due to a complication of bleeding in each participant on admission in labour compared to 24 hours postpartum
Percentage of participants who receive a hysterectomy as a complication of bleeding will be assessed | 24 hours
Percentage of participants who are admitted to the ICU due to complications of bleeding will be assessed | 24 hours
Percentage of participants with fever as a complication of misoprostol administration will be assessed | 24 hours
Percentage of participants with shivering as a complication of misoprostol administration will be assessed (Shivering) | 24 hours
Percentage of participants with nausea as a complication of misoprostol administration will be assessed (Nausea) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rattray Dr Carole, Principal Investigator — University of the West Indies Mona
Locations (1):
- University Hospital of the West Indies, Mona, Kingston, Jamaica